CLINICAL TRIAL: NCT01920412
Title: A Prospective, Non-randomized, Multicenter, Open-label, Non-comparative, First-in-Man Study to Evaluate the Feasibility and Safety of LAmbre Left Atrial Appendage Occluder
Brief Title: Feasibility and Safety Study of LAmbre Left Atrial Appendage Occluder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LA-AP-01
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2013-08

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial fibrillation; Thrombosis; Ischemic stroke; Left atrial appendage occluder; Intervention method
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thrombosis; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Left Atrial Appendage Occluder (Experimental): Adopted non-comparative arm on Left Atrial Appendage Occluder.
  Interventions: Device: LAmbre Left Atrial Appendage(LAA) Occluder

INTERVENTIONS:
Device: LAmbre Left Atrial Appendage(LAA) Occluder — Implanting the LAmbre Left Atrial Appendage Occluder to close the left atrial appendage

SUMMARY:
This study mainly evaluated the feasibility and safety of LAmbre Left Atrial Appendage Occluder which is to prevent ischemic stroke caused by atrial fibrillation(AF).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common arrhythmia, its incidence increases with age. Thrombosis shed off caused by AF is one of the major causes of stroke. Most patients with AF suffer ischemic stroke that the thrombosis was from the left atrial appendage(LAA). The majority of patients with atrial fibrillation, the blood clots come from the left atrial appendage, so close the left atrial appendage can reduce cycle thromboembolism of the patients with AF. Now patients have cardiac surgery and risk at left atrium related thromboembolism, the surgery has been conventional perform the left atrial appendage closed surgery.

However, surgical left atrial appendage ligation is difficult to be completely closed to the left atrial appendage,internal medicine intervention methods of surgical closure the left atrial appendage is relatively simple, minimally invasive, high success rate and is expected to be widely used.

Several versions of LAA occlusion devices have been developed.LAA occluder of Lifetech consists of a umbrella, cover and conveyor; The umbrella composed of multiple umbrella and covered the ePTFE membrane.This study mainly evaluated the feasibility and safety of LAmbre Left Atrial Appendage Occluder! Through the femoral vein puncture; insert inter atrial septum puncture device; puncture a small hole in the atrial septal, delivery sheath is inserted in the femoral vein puncture site and across the atrial septal reach the left atrial appendage, establishment of the channel. Through the built-channel sent the LAA occluder to the left atrial appendage by the delivery cable; The LAA occlude will be fixed in the left atrial appendage, close the entrance of the left atrial appendage meanwhile and block blood flow; then eliminate the risk of blood clots due to atrial fibrillation, prevention stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age;
2. Chronic atrial fibrillation ≥3 months; paroxysmal, persistent or permanent non-valvular AF;
3. CHADS2-VAS score 2 or higher;
4. Patient can understand the trial purpose, voluntarily join this clinical trial with informed consent;
5. Patient voluntarily completes the follow-up and follow-up inspection in accordance with the clinical trials process.

Exclusion Criteria:

* A. Clinical exclusion criteria

  1. Presence of rheumatic, degenerative or congenital valvular heart diseases,
  2. The diameter of left atrial ≥65 mm;
  3. LAA size < 12mm or > 30 mm
  4. Left atrium has been removed;
  5. Heart transplantation patients;
  6. Symptomatic patients with carotid artery disease (such as carotid stenosis ≥ 50%);
  7. Acute myocardial infarction or unstable angina;
  8. Decompensated heart failure (New York Heart Association functional class III-IV);
  9. Recent myocardial infarction (< 3 months);
  10. Patients with an atrial septal defect or received an atrial septal occluder. The patient has an ablation procedure planned within 30 days of potential LAmbre Occluder implant
  11. The patient has a planned cardioversion 30 days post implant of the LAmbre Occluder
  12. Patient who after artificial mechanical heart valve replacement operation;
  13. Uncontrolled Heart rate ≥ 110 beats / min17) History stroke or TIA within 30 days;
  14. Presence of complex aortic plaque(4mm) in ascending aorta;
  15. Cardiac tumors or other malignancy with estimated life expectancy u less than 2 years;
  16. Have thrombocytopenia (platelet 《105 / μl) or anemia（Hb<10g/dl）;
  17. Women who is pregnancy or plan to pregnancy during the trial period;
  18. Presence of active sepsis or endocarditis;
  19. Patient participated in the other trials;
  20. The investigators expect the patient not be able to complete the trial according to requirements.

B. Esophageal ultrasonic exclusion criteria

1. LVEF≤30%;
2. Presence of left atrial appendage thrombus;
3. High risk PFO patients(presence of atrial septal aneurysm);
4. Have obvious mitral valve stenosis (the area of mitral valve≤ 2 cm2);
5. Have obvious and unexplained pericardial effusion(≥4 cm2).
6. Presence of complex aortic plague(≥4 mm) in ascending aorta.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The feasibility end-point | 30 days
  stable device placement in left atrial appendage as assessed by angiography and trans-esophageal(TEE)and successful sealing around the device LAA orifice with the device(jet<3mm in width) as measured by TEE at 30 days after device implant

SECONDARY OUTCOMES:
The composite safety and efficacy end-point | 12 months
  Safety:freedom of major adverse events such as pericardial effusion. Successful closure without evidence of residual shunt and ischemic stroke after 1 year confirmed by trans-esophageal(TEE) and electrocardiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Yat-Yin YY Lam, MD, Principal Investigator — Prince of Wales Hospital, Shatin, Hong Kong; Muhammad Munawar, MD, Principal Investigator — Binawaluya Hospital, Indonesia; Lan Hieu Nguyen, MD, Principal Investigator — Hanoi Heart Hospital, Vietnam; Yan Yao, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Congxin Huang, MD, Principal Investigator — Renmin Hospital of Wuhan University,China
Locations (1):
- Prince of Wales Hospital, Hong Kong, China